CLINICAL TRIAL: NCT05232864
Title: A Three-year, Open-label Extension Study of Subcutaneous Secukinumab to Evaluate the Long-term Efficacy, Safety and Tolerability in Patients With Active Lupus Nephritis
Brief Title: Open-label Extension Study of Efficacy, Safety and Tolerability of Secukinumab in Patients With Active Lupus Nephritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated by sponsor based on a futility analysis of the core study CAIN457Q12301
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457Q12301E1; 2021-005772-19 (EudraCT Number)
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Results first posted 2024-08-30 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Lupus Nephritis
Keywords: Lupus Nephritis; secukinumab (AIN457); estimated glomerular filtration rate; Urine Protein-to-Creatinine Ratio; Standard of Care background therapy
MeSH Terms: conditions — Lupus Nephritis | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Secukinumab (Experimental): Secukinumab 300 mg solution for subcutaneous (s.c.) injection in a 2mL Pre-Filled Syringe (PFS)
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — 300 mg solution for subcutaneous (s.c.) injection in a 2mL Pre-Filled Syringe (PFS)
  Other Names: AIN457

SUMMARY:
The purpose of this open-label extension study was to provide treatment with secukinumab for subjects who completed core study treatment in Study CAIN457Q12301 (NCT04181762), and to obtain further data on long-term efficacy, safety and tolerability of secukinunab in patients with active lupus nephritis (LN).

DETAILED DESCRIPTION:
Investigators used their clinical judgement to decide if it might be beneficial, in terms of overall improvement and response to therapy, for subjects to enter the extension study. The planned total combined duration for the core study and this extension study was five years.

At Week 104 of the core study CAIN457Q12301, eligible subjects who completed the assessments associated with the core study visit subsequently continued in the extension study on the dose of secukinumab 300 mg administered every four weeks.

A total of 31 subjects were enrolled and received secukinumab 300 mg every four weeks until study termination. Recruitment in this study was stopped on 26-May-2023.

This study along with the core study (CAIN457Q12301) were terminated early by Novartis due to futile results of interim analysis 1 of the core study. There were no safety related reasons for early termination of either of the studies.

ELIGIBILITY:
Key inclusion criteria:

* Subject must have both participated in core study and completed the entire treatment period up to and including Week 104 of the core study CAIN457Q12301.
* Subject must be deemed by the investigator to benefit from secukinumab therapy.
* Signed informed consent must be obtained prior to participation in the study.

Key Exclusion criteria:

* Any subject taking other concomitant biologic immunomodulating agent(s) except secukinumab.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
* Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during the entire study or longer if required by locally approved prescribing information (e.g., in European Union (EU) 20 Weeks). Highly effective methods of contraception are recommended due to the known teratogenic effect of SoC (MPA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (16):
- Novartis Investigative Site, Westmead, New South Wales, Australia
- Brazil (2):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Barranquilla, Colombia
- Novartis Investigative Site, Prague, Czechia
- Novartis Investigative Site, Guatemala City, Guatemala
- Japan (2):
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Sendai, Miyagi
- Novartis Investigative Site, Lipa City, Batangas, Philippines
- Portugal (2):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Porto
- Novartis Investigative Site, Piešťany, Slovakia
- Novartis Investigative Site, Seoul, South Korea
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Novartis Investigative Site, Bangkok, Thailand
- Novartis Investigative Site, Ho Chi Minh City, VNM, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Zhao MH, Cons Molina F, Aroca G, Tektonidou MG, Mathur A, Tangadpalli R, Sun R, Martin R, Pellet P, Ngoc Phuong Huynh T. Secukinumab in active lupus nephritis: Results from phase III, randomised, placebo-controlled study (SELUNE) and open-label extension study. Rheumatology (Oxford). 2025 Oct 15:keaf536. doi: 10.1093/rheumatology/keaf536. Online ahead of print. PMID 41092316
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2284

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 18 centers in 13 countries: Australia (1 site), Brazil (2 sites), Colombia (1 site), Czech Republic (2 sites), Guatemala (2 sites), Japan (2 sites), Korea (1 site), Republic of Philippines (1 site), Portugal (2 sites), Slovakia (Slovak Republic) (1 site), Spain (1 site), Thailand (1 site), Vietnam (1 site)
Groups:
- Secukinumab 300 mg: Patients who were on Secukinumab 300 mg in the Core Study (CAIN457Q12301) and continued treatment with Secukinumab 300 mg every four weeks in the Extension Study until study termination notification (maximum treatment exposure during the extension study: 281 days)
- Placebo to Secukinumab 300 mg: Patients who were on Placebo in the Core Study (CAIN457Q12301) and continued treatment with Secukinumab 300 mg every four weeks in the Extension Study until study termination notification (maximum treatment exposure during the extension study: 310 days)
Period: Overall Study
Arm/Group | Secukinumab 300 mg | Placebo to Secukinumab 300 mg
Started (All enrolled subjects were included in the Full Analysis Set and Safety Set) | 16 | 15
Completed | 0 | 0
Not Completed | 16 | 15
Not completed — Adverse Event | 0 | 1
Not completed — Study terminated by sponsor | 16 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab 300 mg | Placebo to Secukinumab 300 mg | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.6 (8.26) | 30.6 (9.83) | 33.2 (9.26)
Age, Customized [Count of Participants; unit: Participants]
  < 30 years | 4 | 7 | 11
  >= 30 years | 12 | 8 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 0 | 6
  Asian | 8 | 8 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 6 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Complete Renal Response (CRR)
Description: Complete Renal Response (CRR) is a composite endpoint defined as:
  * Estimated Glomerular Filtration Rate (eGFR) >= 60 mL/min/1.73 m^2 or no less than 85% of core Baseline values and
  * 24-hour Urine-to-Protein Creatinine Ratio (UPCR) =< 0.5mg/mg
  The glomerular filtration rate was estimated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation based on subject gender, age (years) and serum creatinine (mg/dL). Central laboratory serum creatinine values were used for all renal function data analysis.
  UPCR was determined by a central laboratory by dividing the protein concentration by the creatinine concentration as measured in the urine collected. UPCR was determined using one of the following two types of urine collection, 24-hour urine collection or first morning void urinary sample, both of which were collected in the subjects' home.
Time Frame: Up to 28 weeks: from enrollment in the extension study (Week 104E1) up to Week 132 or Early termination of the Extension Study. Study day is defined with respect to the core study.
Population: Full Analysis Set. Percentages were calculated based on the number of participants with an assessment at the specified time point independently if subject was still on treatment or discontinued from treatment before that timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 300 mg | Placebo to Secukinumab 300 mg
Number analyzed (Participants) | 9 | 9
Participants
  Week 104E1 (Baseline Extension Study) (n = 9, 9) | 4 | 5
  Week 132 (n = 6, 5): number analyzed (Participants) | 6 | 5
  Week 132 (n = 6, 5) | 3 | 5

ADVERSE EVENTS:
Time Frame: On-treatment adverse events and deaths were reported from first dose of study treatment in the Core Study up to 84 days after last dose of study medication in the Extension Study, assessed up to approximately 3 year.
Description: Any sign or symptom that occurred during the conduct of the trial and safety follow-up. The Safety Set included all subjects who received at least one dose of study treatment in the extension trial.
Arm/Group | Secukinumab 300 mg | Placebo to Secukinumab 300 mg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 4/16 | 8/15
Other Adverse Events (participants affected / at risk) | 15/16 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300 mg (N=16) | Placebo to Secukinumab 300 mg (N=15)
Cataract (Eye disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 2
Dengue fever (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0
Endometritis (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bipolar disorder (Psychiatric disorders) | 0 | 1
Lupus nephritis (Renal and urinary disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300 mg (N=16) | Placebo to Secukinumab 300 mg (N=15)
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 2
Amaurosis (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 2
Conjunctivitis allergic (Eye disorders) | 1 | 0
Dark circles under eyes (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 2 | 0
Keratitis (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Anal ulcer (Gastrointestinal disorders) | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1
Gingival hypertrophy (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Chest discomfort (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Injection site bruising (General disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Vaccination site pain (General disorders) | 1 | 0
Cholestatic liver injury (Hepatobiliary disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0
Bacterial vaginosis (Infections and infestations) | 2 | 1
Bacteriuria (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 5 | 7
Cystitis (Infections and infestations) | 0 | 1
Dacryocystitis (Infections and infestations) | 1 | 0
Dermatophytosis of nail (Infections and infestations) | 1 | 1
Fungal foot infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2
Gastrointestinal infection (Infections and infestations) | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 1
Helicobacter infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 5 | 0
Influenza (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2
Onychomycosis (Infections and infestations) | 0 | 1
Oral fungal infection (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 2
Periodontitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 3
Pharyngotonsillitis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 4
Urinary tract infection (Infections and infestations) | 4 | 5
Vaginal infection (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Viral tonsillitis (Infections and infestations) | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Immunisation reaction (Injury, poisoning and procedural complications) | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Folate deficiency (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Metabolic syndrome (Metabolism and nutrition disorders) | 1 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 3 | 0
Intercostal neuralgia (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 2
Irritability (Psychiatric disorders) | 1 | 0
Mood swings (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Lupus nephritis (Renal and urinary disorders) | 0 | 2
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Urine abnormality (Renal and urinary disorders) | 0 | 1
Urine odour abnormal (Renal and urinary disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 | 1
Hydrometra (Reproductive system and breast disorders) | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2
Butterfly rash (Skin and subcutaneous tissue disorders) | 1 | 0
Chloasma (Skin and subcutaneous tissue disorders) | 1 | 0
Chronic cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin plaque (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT05232864/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/64/NCT05232864/SAP_001.pdf